CLINICAL TRIAL: NCT00830882
Title: A Proof of Concept Study to Evaluate the Peak Bronchoprotection Conferred by Single and Chronic Dosing With Levosalbutamol and Racemic Salbutamol in Persistent Asthmatics.
Brief Title: Peak Bronchoprotection Conferred by Levosalbutamol and Racemic Salbutamol
Acronym: NAI007
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Dundee (Other)
Responsible Party: Principal Investigator, Brian J Lipworth, Professor, University of Dundee
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NAI007
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2012-06-12 (Estimated); Status verified 2012-06

CONDITIONS: Asthma
Keywords: asthma; levosalbutamol; genotype; bronchoprotection
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1:levosalbutamol (Experimental): 2 puffs four times a day for 2 weeks
  Interventions: Drug: levosalbutamol
- 2: racemic salbutamol (Active Comparator): 2 puffs four times a day for 2 weeks
  Interventions: Drug: racemic salbutamol
- 3: Placebo (Placebo Comparator): 2 puffs four times a day for 2 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: levosalbutamol — 2 puffs four times a day for 2 weeks
  Arms: 1:levosalbutamol
Drug: racemic salbutamol — 2 puffs four times a day for 2 weeks
  Other Names: ventolin
  Arms: 2: racemic salbutamol
Drug: placebo — 2 puffs four times a day for 2 weeks
  Other Names: placebo to salbutamol
  Arms: 3: Placebo

SUMMARY:
The objective of this study is to compare the peak dose relative bronchoprotection offered by levosalbutamol and racemic salbutamol in mild to moderate asthmatics preselected into two groups on the basis of their beta-2 adrenoreceptor polymorphisms.

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate stable asthmatics on ≤ 2000μg BDP or equivalent
2. Methacholine responsive PC20< 4 mg/ml
3. >1dd change in methacholine PC20 after the administration of racemic Salbutamol.
4. Male or female 18-65
5. Informed Consent
6. Ability to comply with the requirements of the protocol

Exclusion Criteria:

1. Severe asthmatics as defined by an FEV1≤ 60% or PEF variability > 30% or with continual daytime or nocturnal symptoms.
2. The use of oral corticosteroids within the last 3 months.
3. Recent respiratory tract infection (2 months).
4. Significant concomitant respiratory disease such as COPD, CF, ABPA, bronchiectasis and active pulmonary tuberculosis.
5. Any other clinically significant medical condition such as unstable angina, acute myocardial infarction in the preceding 3 months, recent TIA/ CVA,that may endanger the health or safety of the participant, or jeopardise the protocol.
6. Any significant abnormal laboratory result as deemed by the investigators
7. Pregnancy, planned pregnancy or lactation
8. Known or suspected contra-indication to any of the IMP's
9. Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Methacholine challenge | Before and 30 mins after drug administration, and after 2 weeks of chronic treatment

SECONDARY OUTCOMES:
Salbutamol pharmacokinetics | over 30 minutes after drug administration, one day 1 and 14 of a 2 week study period
Spirometry | before and 30 mins after drug administration, at single dose and after 2 weeks chronic dosing
potassium | before and 30 mins after drug administration, at single dose and after 2 weeks chronic dosing

CONTACTS AND LOCATIONS:
Overall Officials: Karine L Clearie, MBBS, MRCP, Principal Investigator — Asthma and Allergy Research Group; Brian J Lipworth, MBchB, Study Director — Asthma and Allergy Research Group
Locations (1):
- Asthma and Allergy Research Group, Dundee, Angus, United Kingdom